CLINICAL TRIAL: NCT06680206
Title: Comparing Patient-Reported Outcomes Between Rimegepant and Triptan Users With Migraine in the United States
Brief Title: Comparison of Patient-reported Outcomes for Rimegepant and Triptans in the 2023 US National Health and Wellness Survey
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4951076; NCT06680206 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-10-21; First posted 2024-11-08 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Migraine
Keywords: Rimegepant; Triptans; Acute treatment of migraine; Survey; Cross-sectional design; National Health and Wellness Survey (NHWS); Patient-reported outcomes; Treatment satisfaction
MeSH Terms: conditions — Migraine Disorders | interventions — rimegepant sulfate; Tryptamines

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: None Retained — No biosamples will be collected in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute treatment of migraine
  Interventions: Drug: Rimegepant; Drug: Triptans

INTERVENTIONS:
Drug: Rimegepant — Rimegepant for acute treatment of migraine
Drug: Triptans — Triptans for acute treatment of migraine

SUMMARY:
This is a cross-sectional study using the cross-sectional 2023 National Health and Wellness Survey (NHWS) data from the US, with a large and nationally representative population (N=75,007).

All data from the NHWS are reported by respondents, who are recruited through an existing, general-purpose, web-based, consumer panel via opt-in e-mails, co-registration with panel partners, e-newsletter campaigns, banner placements, and affiliate networks. All respondents explicitly agree to be a panel member, register with the panel through a unique e-mail address, and complete an in-depth demographic registration profile.

This analysis will focus on respondents who self-report having migraine diagnosed by a physician. Individuals who use rimegepant for acute treatment of migraine will be compared with those who use triptans for acute treatment of migraine. Outcomes of interest include treatment satisfaction, healthcare resource utilization (HCRU), quality of life (QoL), work productivity loss, and migraine-specific disability outcomes.

Inverse probability of treatment weighting (IPTW) will be used to adjust for differences that may exist between rimegepant and triptan users prior to comparing outcomes.

DETAILED DESCRIPTION:
This is a cross-sectional study using the cross-sectional 2023 National Health and Wellness Survey (NHWS) data from the US, with a large and nationally representative population (N=75,007).

All data from the NHWS are reported by respondents, who are recruited through an existing, general-purpose, web-based, consumer panel via opt-in e-mails, co-registration with panel partners, e-newsletter campaigns, banner placements, and affiliate networks. All respondents explicitly agree to be a panel member, register with the panel through a unique e-mail address, and complete an in-depth demographic registration profile.

This analysis will focus on respondents who self-report having migraine diagnosed by a physician. Individuals who use rimegepant for acute treatment of migraine will be compared with those who use triptans for acute treatment of migraine. Outcomes of interest include treatment satisfaction, healthcare resource utilization (HCRU), quality of life (QoL), work productivity loss, and migraine-specific disability outcomes.

Inverse probability of treatment weighting (IPTW) will be used to adjust for differences that may exist between rimegepant and triptan users prior to comparing outcomes.

Additional information is provided in the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Participated in 2023 NHWS in the US
* Consented to the anonymous use of their data for research purpose
* Aged 18 or older
* Self-reported a diagnosis of migraine by physician
* Currently on rimegepant or triptan (via oral route) at the time of the survey

Exclusion Criteria:

- Currently on both rimegepant and triptans at the time of the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will analyze data from 2023 National Health and Wellness Survey (NHWS) in the US. The NHWS is a cross-sectional study intended to be representative of the US population in terms of age, sex, race, and ethnicity.
  This study will focus on NHWS respondents who report a physician diagnosis of migraine.
  This analysis will compare those who report taking rimegepant for acute treatment of migraine and those who report taking triptans for acute treatment of migraine at the time of the survey.
Sampling Method: Non-Probability Sample
Enrollment: 1395 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4951076

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this retrospective observational study, data of participants who used rimegepant or triptans for migraine (diagnosed by physician) in Year 2023, was retrieved from United States National Health and Wellness Survey (NHWS). Retrieved retrospective data was evaluated in approximately 1.41 months (from study start date: 10-Oct-2024 to study completion date: 20-Nov-2024) per objectives of the study.
Groups:
- Rimegepant: Participants with self-reported diagnosis of migraine currently on rimegepant use at the time of survey (NHWS in year 2023) were included. No intervention was administered as part of this study.
- Triptans: Participants with self-reported diagnosis of migraine currently on triptan use at the time of survey (NHWS in year 2023) were included. No intervention was administered as part of this study.
Period: Overall Study
Arm/Group | Rimegepant | Triptans
Started | 137 | 1258
Inverse Probability Treatment Weighting (IPTW) Adjustment (Weighted counts (after IPTW)) | 135 | 1260
Sensitivity Analysis | 105 ('Rimegepant users with less than 12 days of rimegepant use per month') | 1258
Sensitivity Analysis IPTW Adjustment (Weighted counts (after IPTW)) | 103 ('Rimegepant users with less than 12 days of rimegepant use per month') | 1257
Completed | 137 | 1258
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were retrieved and observed in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rimegepant | Triptans | Total
Number analyzed (Participants) | 137 | 1258 | 1395
Age, Customized [Count of Participants; unit: Participants]
  18-29 years | 25 | 178 | 203
  30-39 years | 26 | 185 | 211
  40-49 years | 39 | 249 | 288
  50-59 years | 29 | 282 | 311
  60-69 years | 13 | 248 | 261
  70-79 years | 5 | 108 | 113
  80-89 years | 0 | 8 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 1016 | 1140
  Male | 13 | 242 | 255
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 122 | 140
  Not Hispanic or Latino | 119 | 1136 | 1255
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 12 | 114 | 126
  Race: White | 116 | 1062 | 1178
  Race: Other | 9 | 82 | 91

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants According to Migraine Medication Type (Prescription Drug or Over the Counter [OTC])
Description: Number of participants according to migraine medication type: 1) as prescription drug only, 2) as OTC only or 3) as both prescription drug and OTC based on the use of migraine medication classes is reported in this outcome measure. Analysis was performed using inverse probability treatment weighting (IPTW) method to adjust for confounding by the covariates.
Time Frame: At the time of survey during 1 year of data identification (Year 2023); available retrospective data was evaluated over approximately 1.41 months of this observational study.
Population: Analysis population included all eligible participants whose data were retrieved and observed in the study and were adjusted using IPTW method (pseudo-set); hence, numbers of participants are different here from those presented in participant flow and baseline section.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Participants
  Prescription Drug only | 74 | 682
  Prescription drug and OTC | 61 | 578
  OTC only | 0 | 0
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Test type: Other; p = 0.928, Fisher Exact

2. Primary Outcome: Number of Participants According to Migraine Treatment Type (Acute or Prevention)
Description: Number of participants according to migraine treatment type: 1) acute use only, 2) prevention use only, or 3) both acute and prevention use based on the use of migraine medication classes is reported in this outcome measure. Acute treatments included: triptans, non-steroidal anti-inflammatory drugs (NSAIDs), opioids, barbiturates, ergots, gepants [acute; including Nurtec], ditan, combination analgesics, and other acute treatment; preventive treatment included: anticonvulsants, beta blocker, antidepressant, calcitonin gene-related peptide antibodies monoclonal antibodies (CGRP mAb), botox, and gepant [prevention treatment including Nurtec]). Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Participants
  Acute use only | 0 | 837
  Prevention use only | 0 | 0
  Both Acute and Prevention use | 135 | 423
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Test type: Other; p < 0.001, Fisher Exact

3. Primary Outcome: Total Number of Acute Migraine Agent Drug Classes Used
Description: Total number of distinct acute migraine agent drug classes used by participants is reported as mean in this outcome measure. Acute migraine agents included: triptans, NSAIDs, opioids, barbiturates, ergots, gepants [acute; including Nurtec], ditan, combination analgesics, and other acute treatment. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Drug classes per participant
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Drug classes per participant | 2.1 (1.2) | 2.2 (1.2)
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Test type: Other; p = 0.895, t-test, 2 sided

4. Primary Outcome: Number of Participants According to Number of Acute Migraine Agent Drug Classes Used
Description: Number of participants categorized by the number of distinct acute migraine agent drug classes used is reported in this outcome measure. Categories included 1 drug class, 2 or more drug classes, and 3 or more drug classes. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Participants
  1 drug class | 51 | 431
  2 or more drug classes | 84 | 829
  3 or more drug classes | 40 | 406
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; 1 drug class; Test type: Other; p = 0.463, Chi-squared
Statistical Analysis 2: Comparison: Rimegepant vs Triptans; 2 or more drug classes; Test type: Other; p = 0.463, Chi-squared
Statistical Analysis 3: Comparison: Rimegepant vs Triptans; 3 or more drug classes; Test type: Other; p = 0.644, Chi-squared

5. Primary Outcome: Total Number of Prevention Migraine Agent Drug Classes Used
Description: Preventive migraine agents included: anticonvulsants, beta blocker, antidepressant, CGRP mAb, botox, and gepant [prevention treatment including Nurtec]. Total number of distinct preventive migraine agent drug classes used by participants is reported as mean in this outcome measure. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in the study and were adjusted using IPTW method (pseudo-set); hence, numbers of participants are different here from those presented in participant flow and baseline section. The analysis was performed on all participants reported under Overall Number of Participants Analyzed.
Measure: Mean (Standard Deviation); unit: Drug classes per participant
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Drug classes per participant | 1.5 (0.7) | 0.5 (0.8)
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Test type: Other; p < 0.001, t-test, 2 sided

6. Primary Outcome: Number of Participants According to Number of Prevention Migraine Agent Drug Classes Used
Description: Number of participants categorized by the number of distinct prescription preventive migraine agent drug classes used reported in this outcome measure. Categories included use of 1 drug class, 2 or more drug classes, and 3 or more drug classes. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Participants
  1 drug class | 79 | 297
  2 or more drug classes | 56 | 126
  3 or more drug classes | 12 | 25
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; 1 drug class; Test type: Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Rimegepant vs Triptans; 2 or more drug classes; Test type: Other; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: Rimegepant vs Triptans; 3 or more drug classes; Test type: Other; p < 0.001, Chi-squared

7. Primary Outcome: Number of Participants According to Current Migraine Treatments
Description: Number of participants according to current migraine treatments on drug classes including: Nurtec (rimegepant) only, acute agents, triptans, NSAIDs, opioids, barbiturates, ergots, gepants [acute; including Nurtec], ditan, combination analgesics, and other acute treatment (aspirin lysine/metoclopramide hydrochloride monohydrate or indometacin/caffeine/prochlorperazine), prevention agents (anticonvulsants, beta-blocker, antidepressant, CGRP mAb, botox, and gepant) are reported in this outcome measure. One participant could receive more than one migraine treatment. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Participants
  Nurtec (rimegepant) only | 135 | 0
  Acute agents | 135 | 1259
  Triptans | 0 | 1260
  NSAIDs | 22 | 187
  Opioids | 10 | 132
  Barbiturates | 6 | 96
  Ergots | 4 | 35
  Gepants (acute; including Nurtec) | 135 | 33
  Ditan | 0 | 3
  Combination analgesics | 18 | 206
  Other (acute treatment) | 2 | 20
  Prevention agents | 135 | 423
  Anticonvulsants | 18 | 191
  Beta blocker | 2 | 45
  Antidepressant | 8 | 53
  CGRP mAb | 28 | 188
  Botox | 15 | 76
  Gepant (prevention treatment including Nurtec) | 135 | 29
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Nurtec (rimegepant) only; Test type: Other; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Rimegepant vs Triptans; Triptans; Test type: Other; p < 0.001, Fisher Exact
Statistical Analysis 3: Comparison: Rimegepant vs Triptans; NSAIDs; Test type: Other; p = 0.746, Chi-squared
Statistical Analysis 4: Comparison: Rimegepant vs Triptans; Opioids; Test type: Other; p = 0.319, Chi-squared
Statistical Analysis 5: Comparison: Rimegepant vs Triptans; Barbiturates; Test type: Other; p = 0.223, Fisher Exact
Statistical Analysis 6: Comparison: Rimegepant vs Triptans; Ergots; Test type: Other; p = 0.791, Fisher Exact
Statistical Analysis 7: Comparison: Rimegepant vs Triptans; Gepants (acute; including Nurtec); Test type: Other; p < 0.001, Chi-squared
Statistical Analysis 8: Comparison: Rimegepant vs Triptans; Ditan; Test type: Other; p = 1.000, Fisher Exact
Statistical Analysis 9: Comparison: Rimegepant vs Triptans; Combination analgesics; Test type: Other; p = 0.447, Chi-squared
Statistical Analysis 10: Comparison: Rimegepant vs Triptans; Other (acute treatment); Test type: Other; p = 1.000, Fisher Exact
Statistical Analysis 11: Comparison: Rimegepant vs Triptans; Prevention agents; Test type: Other; p < 0.001, Chi-squared
Statistical Analysis 12: Comparison: Rimegepant vs Triptans; Anticonvulsants; Test type: Other; p = 0.661, Chi-squared
Statistical Analysis 13: Comparison: Rimegepant vs Triptans; Beta blocker; Test type: Other; p = 0.315, Fisher Exact
Statistical Analysis 14: Comparison: Rimegepant vs Triptans; Antidepressant; Test type: Other; p = 0.377, Chi-squared
Statistical Analysis 15: Comparison: Rimegepant vs Triptans; CGRP mAb; Test type: Other; p = 0.093, Chi-squared
Statistical Analysis 16: Comparison: Rimegepant vs Triptans; Botox; Test type: Other; p = 0.041, Chi-squared
Statistical Analysis 17: Comparison: Rimegepant vs Triptans; Gepant (prevention treatment including Nurtec); Test type: Other; p < 0.001, Chi-squared

8. Primary Outcome: Number of Participants According to Treatment Satisfaction of Migraine Drug Class
Description: Number of participants according to treatment satisfaction for the migraine drug classes including: acute agents, NSAIDs, opioids, barbiturates, ergots, gepants (acute), ditans, combination analgesics, other, prevention agents, anticonvulsants, beta blockers, antidepressants, CGRPs mAb, botox, and gepant reported in this outcome measure. Treatment satisfaction for each of the migraine drug class was categorized as: extremely dissatisfied, very dissatisfied, somewhat dissatisfied, neither dissatisfied nor satisfied, somewhat satisfied, very satisfied, extremely satisfied. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in the study and were adjusted using IPTW method (pseudo-set); hence, numbers of participants are different here from those presented in participant flow and baseline section. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Participants
  Current migraine satisfactions - Acute agents: number analyzed (Participants) | 135 | 1259
  Current migraine satisfactions - Acute agents: Extremely dissatisfied | 3 | 97
  Current migraine satisfactions - Acute agents: Very dissatisfied | 3 | 45
  Current migraine satisfactions - Acute agents: Somewhat dissatisfied | 6 | 92
  Current migraine satisfactions - Acute agents: Neither dissatisfied nor satisfied | 14 | 145
  Current migraine satisfactions - Acute agents: Somewhat satisfied | 36 | 351
  Current migraine satisfactions - Acute agents: Very satisfied | 42 | 341
  Current migraine satisfactions - Acute agents: Extremely satisfied | 31 | 188
  Current migraine satisfactions - NSAIDs: number analyzed (Participants) | 22 | 187
  Current migraine satisfactions - NSAIDs: Extremely dissatisfied | 0 | 15
  Current migraine satisfactions - NSAIDs: Very dissatisfied | 1 | 13
  Current migraine satisfactions - NSAIDs: Somewhat dissatisfied | 2 | 8
  Current migraine satisfactions - NSAIDs: Neither dissatisfied nor satisfied | 4 | 24
  Current migraine satisfactions - NSAIDs: Somewhat satisfied | 10 | 65
  Current migraine satisfactions - NSAIDs: Very satisfied | 3 | 45
  Current migraine satisfactions - NSAIDs: Extremely satisfied | 2 | 17
  Current migraine satisfactions - Opioids: number analyzed (Participants) | 10 | 132
  Current migraine satisfactions - Opioids: Extremely dissatisfied | 0 | 22
  Current migraine satisfactions - Opioids: Very dissatisfied | 0 | 13
  Current migraine satisfactions - Opioids: Somewhat dissatisfied | 2 | 5
  Current migraine satisfactions - Opioids: Neither dissatisfied nor satisfied | 3 | 45
  Current migraine satisfactions - Opioids: Somewhat satisfied | 2 | 23
  Current migraine satisfactions - Opioids: Very satisfied | 2 | 17
  Current migraine satisfactions - Opioids: Extremely satisfied | 1 | 7
  Current migraine satisfactions - Barbiturates: number analyzed (Participants) | 6 | 96
  Current migraine satisfactions - Barbiturates: Extremely dissatisfied | 0 | 6
  Current migraine satisfactions - Barbiturates: Very dissatisfied | 1 | 40
  Current migraine satisfactions - Barbiturates: Somewhat dissatisfied | 0 | 11
  Current migraine satisfactions - Barbiturates: Neither dissatisfied nor satisfied | 2 | 10
  Current migraine satisfactions - Barbiturates: Somewhat satisfied | 2 | 18
  Current migraine satisfactions - Barbiturates: Very satisfied | 1 | 9
  Current migraine satisfactions - Barbiturates: Extremely satisfied | 0 | 2
  Current migraine satisfactions - Ergots: number analyzed (Participants) | 4 | 35
  Current migraine satisfactions - Ergots: Extremely dissatisfied | 1 | 0
  Current migraine satisfactions - Ergots: Very dissatisfied | 0 | 2
  Current migraine satisfactions - Ergots: Somewhat dissatisfied | 1 | 0
  Current migraine satisfactions - Ergots: Neither dissatisfied nor satisfied | 0 | 0
  Current migraine satisfactions - Ergots: Somewhat satisfied | 0 | 1
  Current migraine satisfactions - Ergots: Very satisfied | 2 | 1
  Current migraine satisfactions - Ergots: Extremely satisfied | 0 | 31
  Current migraine satisfactions - Gepants (acute; including Nurtec): number analyzed (Participants) | 135 | 33
  Current migraine satisfactions - Gepants (acute; including Nurtec): Extremely dissatisfied | 2 | 6
  Current migraine satisfactions - Gepants (acute; including Nurtec): Very dissatisfied | 1 | 0
  Current migraine satisfactions - Gepants (acute; including Nurtec): Somewhat dissatisfied | 4 | 0
  Current migraine satisfactions - Gepants (acute; including Nurtec): Neither dissatisfied nor satisfied | 6 | 3
  Current migraine satisfactions - Gepants (acute; including Nurtec): Somewhat satisfied | 32 | 14
  Current migraine satisfactions - Gepants (acute; including Nurtec): Very satisfied | 52 | 8
  Current migraine satisfactions - Gepants (acute; including Nurtec): Extremely satisfied | 38 | 2
  Current migraine satisfactions - Ditans: number analyzed (Participants) | 0 | 3
  Current migraine satisfactions - Ditans: Extremely dissatisfied | 0 | 0
  Current migraine satisfactions - Ditans: Very dissatisfied | 0 | 0
  Current migraine satisfactions - Ditans: Somewhat dissatisfied | 0 | 0
  Current migraine satisfactions - Ditans: Neither dissatisfied nor satisfied | 0 | 0
  Current migraine satisfactions - Ditans: Somewhat satisfied | 0 | 2
  Current migraine satisfactions - Ditans: Very satisfied | 0 | 1
  Current migraine satisfactions - Ditans: Extremely satisfied | 0 | 0
  Current migraine satisfactions - Combination Analgesics: number analyzed (Participants) | 18 | 206
  Current migraine satisfactions - Combination Analgesics: Extremely dissatisfied | 0 | 11
  Current migraine satisfactions - Combination Analgesics: Very dissatisfied | 1 | 13
  Current migraine satisfactions - Combination Analgesics: Somewhat dissatisfied | 2 | 21
  Current migraine satisfactions - Combination Analgesics: Neither dissatisfied nor satisfied | 4 | 40
  Current migraine satisfactions - Combination Analgesics: Somewhat satisfied | 6 | 71
  Current migraine satisfactions - Combination Analgesics: Very satisfied | 5 | 30
  Current migraine satisfactions - Combination Analgesics: Extremely satisfied | 0 | 20
  Current migraine satisfactions - Other (Acute treatment): number analyzed (Participants) | 2 | 20
  Current migraine satisfactions - Other (Acute treatment): Extremely dissatisfied | 0 | 6
  Current migraine satisfactions - Other (Acute treatment): Very dissatisfied | 0 | 0
  Current migraine satisfactions - Other (Acute treatment): Somewhat dissatisfied | 0 | 0
  Current migraine satisfactions - Other (Acute treatment): Neither dissatisfied nor satisfied | 0 | 7
  Current migraine satisfactions - Other (Acute treatment): Somewhat satisfied | 0 | 2
  Current migraine satisfactions - Other (Acute treatment): Very satisfied | 0 | 5
  Current migraine satisfactions - Other (Acute treatment): Extremely satisfied | 2 | 0
  Current migraine satisfactions - Prevention agents: number analyzed (Participants) | 135 | 423
  Current migraine satisfactions - Prevention agents: Extremely dissatisfied | 2 | 28
  Current migraine satisfactions - Prevention agents: Very dissatisfied | 1 | 12
  Current migraine satisfactions - Prevention agents: Somewhat dissatisfied | 9 | 21
  Current migraine satisfactions - Prevention agents: Neither dissatisfied nor satisfied | 14 | 106
  Current migraine satisfactions - Prevention agents: Somewhat satisfied | 29 | 107
  Current migraine satisfactions - Prevention agents: Very satisfied | 47 | 85
  Current migraine satisfactions - Prevention agents: Extremely satisfied | 33 | 64
  Current migraine satisfactions - Anticonvulsants: number analyzed (Participants) | 18 | 191
  Current migraine satisfactions - Anticonvulsants: Extremely dissatisfied | 0 | 25
  Current migraine satisfactions - Anticonvulsants: Very dissatisfied | 0 | 4
  Current migraine satisfactions - Anticonvulsants: Somewhat dissatisfied | 2 | 11
  Current migraine satisfactions - Anticonvulsants: Neither dissatisfied nor satisfied | 4 | 38
  Current migraine satisfactions - Anticonvulsants: Somewhat satisfied | 3 | 47
  Current migraine satisfactions - Anticonvulsants: Very satisfied | 4 | 43
  Current migraine satisfactions - Anticonvulsants: Extremely satisfied | 5 | 23
  Current migraine satisfactions - Beta-blockers: number analyzed (Participants) | 2 | 45
  Current migraine satisfactions - Beta-blockers: Extremely dissatisfied | 0 | 7
  Current migraine satisfactions - Beta-blockers: Very dissatisfied | 0 | 6
  Current migraine satisfactions - Beta-blockers: Somewhat dissatisfied | 0 | 2
  Current migraine satisfactions - Beta-blockers: Neither dissatisfied nor satisfied | 0 | 2
  Current migraine satisfactions - Beta-blockers: Somewhat satisfied | 1 | 11
  Current migraine satisfactions - Beta-blockers: Very satisfied | 1 | 6
  Current migraine satisfactions - Beta-blockers: Extremely satisfied | 0 | 11
  Current migraine satisfactions - Antidepressants: number analyzed (Participants) | 8 | 53
  Current migraine satisfactions - Antidepressants: Extremely dissatisfied | 0 | 7
  Current migraine satisfactions - Antidepressants: Very dissatisfied | 0 | 0
  Current migraine satisfactions - Antidepressants: Somewhat dissatisfied | 2 | 0
  Current migraine satisfactions - Antidepressants: Neither dissatisfied nor satisfied | 2 | 17
  Current migraine satisfactions - Antidepressants: Somewhat satisfied | 1 | 11
  Current migraine satisfactions - Antidepressants: Very satisfied | 3 | 13
  Current migraine satisfactions - Antidepressants: Extremely satisfied | 0 | 5
  Current migraine satisfactions - CGRPs mAb: number analyzed (Participants) | 28 | 188
  Current migraine satisfactions - CGRPs mAb: Extremely dissatisfied | 1 | 2
  Current migraine satisfactions - CGRPs mAb: Very dissatisfied | 0 | 1
  Current migraine satisfactions - CGRPs mAb: Somewhat dissatisfied | 0 | 4
  Current migraine satisfactions - CGRPs mAb: Neither dissatisfied nor satisfied | 1 | 51
  Current migraine satisfactions - CGRPs mAb: Somewhat satisfied | 5 | 47
  Current migraine satisfactions - CGRPs mAb: Very satisfied | 9 | 34
  Current migraine satisfactions - CGRPs mAb: Extremely satisfied | 12 | 49
  Current migraine satisfactions - Botox: number analyzed (Participants) | 15 | 76
  Current migraine satisfactions - Botox: Extremely dissatisfied | 0 | 0
  Current migraine satisfactions - Botox: Very dissatisfied | 1 | 1
  Current migraine satisfactions - Botox: Somewhat dissatisfied | 1 | 0
  Current migraine satisfactions - Botox: Neither dissatisfied nor satisfied | 1 | 3
  Current migraine satisfactions - Botox: Somewhat satisfied | 3 | 33
  Current migraine satisfactions - Botox: Very satisfied | 7 | 23
  Current migraine satisfactions - Botox: Extremely satisfied | 2 | 16
  Current migraine satisfactions - Gepant (prevention treatment including Nurtec): number analyzed (Participants) | 135 | 29
  Current migraine satisfactions - Gepant (prevention treatment including Nurtec): Extremely dissatisfied | 1 | 0
  Current migraine satisfactions - Gepant (prevention treatment including Nurtec): Very dissatisfied | 1 | 0
  Current migraine satisfactions - Gepant (prevention treatment including Nurtec): Somewhat dissatisfied | 4 | 4
  Current migraine satisfactions - Gepant (prevention treatment including Nurtec): Neither dissatisfied nor satisfied | 7 | 1
  Current migraine satisfactions - Gepant (prevention treatment including Nurtec): Somewhat satisfied | 32 | 12
  Current migraine satisfactions - Gepant (prevention treatment including Nurtec): Very satisfied | 51 | 9
  Current migraine satisfactions - Gepant (prevention treatment including Nurtec): Extremely satisfied | 39 | 3
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Current migraine satisfactions - Acute agents; Test type: Other; p = 0.030, Fisher Exact
Statistical Analysis 2: Comparison: Rimegepant vs Triptans; Current migraine satisfactions - NSAIDs; Test type: Other; p = 0.518, Fisher Exact
Statistical Analysis 3: Comparison: Rimegepant vs Triptans; Current migraine satisfactions - Opioids; Test type: Other; p = 0.184, Fisher Exact
Statistical Analysis 4: Comparison: Rimegepant vs Triptans; Current migraine satisfactions - Barbiturates; Test type: Other; p = 0.333, Fisher Exact
Statistical Analysis 5: Comparison: Rimegepant vs Triptans; Current migraine satisfactions - Ergots; Test type: Other; p < 0.001, Fisher Exact
Statistical Analysis 6: Comparison: Rimegepant vs Triptans; Current migraine satisfactions - Gepants (acute; including Nurtec); Test type: Other; p < 0.001, Fisher Exact
Statistical Analysis 7: Comparison: Rimegepant vs Triptans; Current migraine satisfactions - Combination Analgesics; Test type: Other; p = 0.680, Fisher Exact
Statistical Analysis 8: Comparison: Rimegepant vs Triptans; Current migraine satisfactions - Other (Acute treatment); Test type: Other; p = 0.011, Fisher Exact
Statistical Analysis 9: Comparison: Rimegepant vs Triptans; Current migraine satisfactions - Prevention agents; Test type: Other; p < 0.001, Fisher Exact
Statistical Analysis 10: Comparison: Rimegepant vs Triptans; Current migraine satisfactions - Anticonvulsants; Test type: Other; p = 0.314, Fisher Exact
Statistical Analysis 11: Comparison: Rimegepant vs Triptans; Current migraine satisfactions - Beta-blockers; Test type: Other; p = 0.890, Fisher Exact
Statistical Analysis 12: Comparison: Rimegepant vs Triptans; Current migraine satisfactions - Antidepressants; Test type: Other; p = 0.055, Fisher Exact
Statistical Analysis 13: Comparison: Rimegepant vs Triptans; Current migraine satisfactions - CGRPs mAb; Test type: Other; p = 0.016, Fisher Exact
Statistical Analysis 14: Comparison: Rimegepant vs Triptans; Current migraine satisfactions - Botox; Test type: Other; p = 0.079, Fisher Exact
Statistical Analysis 15: Comparison: Rimegepant vs Triptans; Current migraine satisfactions - Gepant (prevention treatment including Nurtec); Test type: Other; p = 0.079, Fisher Exact

9. Primary Outcome: Number of Participants According to Current Migraine Treatments on OTC Class
Description: Participants were categorized based on current use of OTC migraine treatments, including analgesics (acetaminophen only), analgesics (combination), NSAIDs, and other OTCs.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in the study and were adjusted using IPTW method (pseudo-set); hence, numbers of participants are different here from those presented in participant flow and baseline section. Analysis was performed on all participants reported under "Overall Number of Participants Analyzed".
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Participants
  Analgesics (acetaminophen only) | 34 | 198
  Analgesics (Combination) | 28 | 221
  NSAIDs | 32 | 320
  Other | 0 | 4
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Analgesics (acetaminophen only); Test type: Other; p = 0.011, Chi-squared
Statistical Analysis 2: Comparison: Rimegepant vs Triptans; Analgesics (Combination); Test type: Other; p = 0.421, Chi-squared
Statistical Analysis 3: Comparison: Rimegepant vs Triptans; NSAIDs; Test type: Other; p = 0.636, Chi-squared
Statistical Analysis 4: Comparison: Rimegepant vs Triptans; Other; Test type: Other; p = 1.000, Fisher Exact

10. Primary Outcome: Number of Participants According to Treatment Satisfaction of Analgesics (Acetaminophen Only)
Description: Number of participants according to treatment satisfaction for analgesics (acetaminophen only) is reported in this outcome measure. Treatment satisfaction was categorized as: extremely dissatisfied, very dissatisfied, somewhat dissatisfied, neither dissatisfied nor satisfied, somewhat satisfied, very satisfied, extremely satisfied. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in the study and were adjusted using IPTW method (pseudo-set); hence, numbers of participants are different here from those presented in participant flow and baseline section. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 34 | 198
Participants
  Extremely dissatisfied | 3 | 13
  Very dissatisfied | 2 | 3
  Somewhat dissatisfied | 6 | 13
  Neither dissatisfied nor satisfied | 10 | 44
  Somewhat satisfied | 12 | 93
  Very satisfied | 1 | 24
  Extremely satisfied | 0 | 8
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Test type: Other; p = 0.050, Fisher Exact

11. Primary Outcome: Number of Participants According to Treatment Satisfaction to Rimegepant or Triptans
Description: Number of participants according to treatment satisfaction for rimegepant or triptans is reported in this outcome measure. Treatment satisfaction was categorized as: extremely dissatisfied, very dissatisfied, somewhat dissatisfied, neither dissatisfied nor satisfied, somewhat satisfied, very satisfied, extremely satisfied. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Participants
  Extremely dissatisfied | 1 | 74
  Very dissatisfied | 1 | 46
  Somewhat dissatisfied | 4 | 69
  Neither dissatisfied nor satisfied | 7 | 101
  Somewhat satisfied | 32 | 333
  Very satisfied | 51 | 389
  Extremely satisfied | 39 | 248
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Test type: Other; p = 0.002, Fisher Exact

12. Primary Outcome: Research and Development (RAND-36) Physical Component Score, Mental Component Score and Global Health Score - Primary Analysis
Description: RAND-36=standardized survey evaluating 8 domains of functional health and well-being: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health. Score for each of the 8 domains were scaled from 0=worst condition to 100=best condition, higher scores indicated better health status. These 8 domains were summarized as summary scores: physical component scores (derived from physical functioning, role physical, bodily pain, general health), mental component scores (derived from social functioning, role emotional mental health and vitality) and global health composite score (derived from physical and mental component scores). Each of the summary scores were standardized to a T-score with mean=50 and SD=10. Scores ranged from 0 to 100, where 0 (worst condition) to 100 (best condition), where higher scores represent better health status. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Units on a scale
  Mental summary composite T score | 38.2 (12) | 37.1 (12.6)
  Physical summary composite T score | 39.5 (12) | 39.8 (11.9)
  Global health composite T score | 37.2 (12.4) | 36.7 (12.7)
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Mental summary composite T score; Test type: Other; p = 0.308, t-test, 2 sided
Statistical Analysis 2: Comparison: Rimegepant vs Triptans; Physical summary composite T score; Test type: Other; p = 0.781, t-test, 2 sided
Statistical Analysis 3: Comparison: Rimegepant vs Triptans; Global health composite T score; Test type: Other; p = 0.637, t-test, 2 sided

13. Primary Outcome: European Quality of Life 5 Dimensions 5 Level (EQ-5D-5L) Index Score - Primary Analysis
Description: EQ-5D-5L is participant completed questionnaire that consisted of two components: a five-item health state profile and visual analog scale (VAS). EQ-5D health state profile had 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension had 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems and 5= extreme problems. Responses to 5 dimensions comprised health state/a single utility index value. E.g. if a participant responds "no problems" for each 5 dimensions, then health state was coded as "11111" with a predefined index value to it. Every health state (coded as combination of responses) had unique predefined utility index value assigned to it per US value sets, by EuroQol. Index scores ranged from -0.59 to 1; where 1 =best possible health state. Negative values= health states perceived as worse than dead, (death=0). Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Units on a scale | 0.7 (0.2) | 0.7 (0.2)
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Test type: Other; p = 0.372, t-test, 2 sided

14. Primary Outcome: EQ-5D-5L Visual Analog Scale (VAS) Score - Primary Analysis
Description: The EQ-5D-5L is a participant completed questionnaire that consisted of two components: a five-item health state profile and a VAS. EQ-5D VAS was used to record participant's rating for his/her current health state on a vertical VAS with scores ranging from 0 to 100, where 0 = worst imaginable health state and 100 = best imaginable health state. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Units on a scale | 66.5 (21.8) | 66.8 (20.6)
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Test type: Other; p = 0.878, t-test, 2 sided

15. Primary Outcome: Percentage of Work Time Missed in Past 7 Days Based on Work Productivity and Activity Impairment - General Health (WPAI-GH) Questionnaire- Primary Analysis
Description: The WPAI is a standardized Patient reported outcome (PRO) that assessed the previous 7 days of completing the questionnaire. WPAI:GH is a self-reported measure of work productivity and impairment, which had four scores: absenteeism (work time missed); presenteeism (impairment at work/reduced on the job effectiveness); work productivity loss (overall work impairment/absenteeism plus presenteeism); and total activity impairment. The scores for percentage of work time missed ranged from 0 (no impairment/high productivity) to-100% (total loss of work productivity) with higher score indicating greater impairment and less productivity. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: 7 days before the survey was taken, during 1 year of data identification (Year 2023); available retrospective data was evaluated over approximately 1.41 months of this observational study.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage work time missed
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Percentage work time missed | 7.1 (17.1) | 9.6 (19.9)
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Test type: Other; p = 0.25, t-test, 2 sided

16. Primary Outcome: Percentage Impairment Experienced While at Work in Past 7 Days Based on WPAI-GH Questionnaire- Primary Analysis
Description: The WPAI is a standardized PRO that assessed the previous 7 days of completing the questionnaire. WPAI:GH is a self-reported measure of work productivity and impairment, which had four scores: absenteeism (work time missed); presenteeism (impairment at work/reduced on the job effectiveness); work productivity loss (overall work impairment/absenteeism plus presenteeism); and total activity impairment. The scores for percentage impairment experienced ranged from 0 (no impairment/high productivity/high impairment) to 100% (total loss of work productivity) with higher score indicating greater impairment and less productivity. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage impairment
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Percentage impairment | 29.4 (26.2) | 27.6 (25.4)
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Test type: Other; p = 0.582, t-test, 2 sided

17. Primary Outcome: Percentage Overall Work Impairment in Past 7 Days Based on WPAI-GH Questionnaire- Primary Analysis
Description: The WPAI is a standardized PRO that assessed the previous 7 days of completing the questionnaire. WPAI:GH is a self-reported measure of work productivity and impairment, which had four scores: absenteeism (work time missed); presenteeism (impairment at work/reduced on the job effectiveness); work productivity loss (overall work impairment/absenteeism plus presenteeism); and total activity impairment. The scores for percentage overall work impairment experienced ranged from 0 (no impairment/high productivity/high impairment) to 100% (total loss of work productivity/high impairment) with higher score indicating greater impairment and less productivity. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage work impairment
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Percentage work impairment | 31.6 (28.1) | 31.1 (28.5)
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Test type: Other; p = 0.898, t-test, 2 sided

18. Primary Outcome: Percentage Total Activity Impairment in Past 7 Days Based on WPAI-GH Questionnaire- Primary Analysis
Description: The WPAI is a standardized PRO that assessed the previous 7 days of completing the questionnaire. WPAI:GH is a self-reported measure of work productivity and impairment, which had four scores: absenteeism (work time missed); presenteeism (impairment at work/reduced on the job effectiveness); work productivity loss (overall work impairment/absenteeism plus presenteeism); and total activity impairment. The scores for percentage of total activity impairment ranged from 0 (no impairment/high productivity) to 100% (total loss of work productivity/high impairment) with higher score indicating greater impairment and less productivity. In this outcome measure, percentage total activity impairment among total population, employed, unemployed and disabled is reported. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 15
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage activity impairment
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Percentage activity impairment
  Total activity impairment | 41.3 (29.3) | 37.6 (28.6)
  Activity impairment among employed: number analyzed (Participants) | 78 | 761
  Activity impairment among employed | 31.8 (26.4) | 31.1 (26.5)
  Activity impairment among unemployed: number analyzed (Participants) | 41 | 393
  Activity impairment among unemployed | 48.8 (27.4) | 41.6 (27.9)
  Activity impairment among disabled: number analyzed (Participants) | 16 | 106
  Activity impairment among disabled | 70 (23.9) | 69.4 (21)
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Total Activity impairment; Test type: Other; p = 0.157, t-test, 2 sided
Statistical Analysis 2: Comparison: Rimegepant vs Triptans; Activity impairment among employed; Test type: Other; p = 0.825, t-test, 2 sided
Statistical Analysis 3: Comparison: Rimegepant vs Triptans; Activity impairment among unemployed; Test type: Other; p = 0.117, t-test, 2 sided
Statistical Analysis 4: Comparison: Rimegepant vs Triptans; Activity impairment among disabled; Test type: Other; p = 0.921, t-test, 2 sided

19. Primary Outcome: Migraine Disability Assessment Scale (MIDAS) Total Score and Individual Item Scores- Primary Analysis
Description: MIDAS is a retrospective, self-administered, 7-item questionnaire that measured headache-related disability as lost time due to headache from paid work or school, household work, and non-work activities. Participants provided the number of missed work or school days (MIDAS Item 1); missed household chores days (MIDAS Item 2); missed social or leisure activity days (MIDAS Item 3); and days with productivity loss at work or school (MIDAS Item 4), days with productivity loss in household work (MIDAS Item 5), frequency of headaches (MIDAS Item 6) and the intensity of the headache pain (MIDAS Item 7). The score ranged from 0 (no disability) to 90 (maximum disability) for each of individual item scores. The 5 item scores (Item 1 to Item 5) were summed to compute the MIDAS total score ranging from 0 (no disability) to 450 (maximum disability). Lower scores indicate less headache-related disability. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: 3 months before the survey was taken, during 1 year of data identification (Year 2023); available retrospective data was evaluated over approximately 1.41 months of this observational study.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Units on a scale
  MIDAS (Total score) | 32.1 (40.8) | 26.8 (36)
  MIDAS Item 1 (MGMIDAS1) | 2.0 (5.5) | 2.1 (6.1)
  MIDAS Item 2 (MGMIDAS2) | 6.8 (12.2) | 4.9 (9.6)
  MIDAS Item 3 (MGMIDAS3) | 9.9 (13.5) | 7.2 (9.7)
  MIDAS Item 4 (MGMIDAS4) | 8.8 (11.6) | 7.6 (10.4)
  MIDAS Item 5 (MGMIDAS5) | 4.7 (8.3) | 5.0 (10.4)
  MIDAS Item 6 (MGMIDAS6) | 21.8 (23.0) | 16.6 (19.8)
  MIDAS Item 7 (MGMIDAS7) | 6.9 (1.8) | 6.9 (1.9)
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; MIDAS (Total score); Test type: Other; p = 0.146, t-test, 2 sided
Statistical Analysis 2: Comparison: Rimegepant vs Triptans; MIDAS Item 1 (MGMIDAS1); Test type: Other; p = 0.741, t-test, 2 sided
Statistical Analysis 3: Comparison: Rimegepant vs Triptans; MIDAS Item 2 (MGMIDAS2); Test type: Other; p = 0.080, t-test, 2 sided
Statistical Analysis 4: Comparison: Rimegepant vs Triptans; MIDAS Item 3 (MGMIDAS3); Test type: Other; p = 0.026, t-test, 2 sided
Statistical Analysis 5: Comparison: Rimegepant vs Triptans; MIDAS Item 4 (MGMIDAS4); Test type: Other; p = 0.254, t-test, 2 sided
Statistical Analysis 6: Comparison: Rimegepant vs Triptans; MIDAS Item 5 (MGMIDAS5); Test type: Other; p = 0.723, t-test, 2 sided
Statistical Analysis 7: Comparison: Rimegepant vs Triptans; MIDAS Item 6 (MGMIDAS6); Test type: Other; p = 0.012, t-test, 2 sided
Statistical Analysis 8: Comparison: Rimegepant vs Triptans; MIDAS Item 7 (MGMIDAS7); Test type: Other; p = 0.807, t-test, 2 sided

20. Primary Outcome: Number of Participants According to MIDAS Grade- Primary Analysis
Description: MIDAS is a retrospective, self-administered, 7-item questionnaire that measured headache-related disability as days with lost time or productivity due to headache from paid work or school, household work, and non-work activities. Participants were categorized according to MIDAS scores as Grade I = Little or No Disability (Score: 0-5), Grade II= Mild Disability (Score: 6-10), Grade III = Moderate Disability (Score: 11-20), Grade IV =severe disability (Score: >=21). Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 19
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Participants
  MIDAS Grade I | 36 | 363
  MIDAS Grade II | 20 | 138
  MIDAS Grade III | 25 | 238
  MIDAS Grade IV | 54 | 521
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; MIDAS Grade I to Grade IV; Test type: Other; p = 0.601, Chi-squared

21. Primary Outcome: Number of Participants With Emergency Room (ER) Visits in Past 6 Months- Primary Analysis
Description: Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: 6 months before the survey was taken, during 1 year of data identification (Year 2023); available retrospective data was evaluated over approximately 1.41 months of this observational study.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Participants | 36 | 334
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Test type: Other; p = 1, Chi-squared

22. Primary Outcome: Number of ER Visits in Past 6 Months- Primary Analysis
Description: Number of ER visits within the last six months due to any cause among those who had at least 1 ER visit reported as mean in this outcome measure. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 21
Population: Analysis population included all eligible participants whose data were retrieved and observed in the study and were adjusted using IPTW method (pseudo-set); hence, numbers of participants are different here from those presented in participant flow and baseline section. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ER visits
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 36 | 334
ER visits | 0.5 (1.1) | 0.5 (1.4)
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Test type: Other; p = 0.688, t-test, 2 sided

23. Primary Outcome: Number of Participants With Hospitalizations in Past 6 Months- Primary Analysis
Description: Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Participants | 15 | 147
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Test type: Other; p = 0.96, Chi-squared

24. Primary Outcome: Mean Number of Hospitalizations in Past 6 Months - Primary Analysis
Description: Mean number of hospitalizations within the last six months due to any cause among those who had at least 1 hospitalization is reported in this outcome measure. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 21
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Hospitalizations
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 15 | 147
Hospitalizations | 1.5 (1.1) | 2.5 (6.6)
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Test type: Other; p = 0.115, t-test, 2 sided

25. Primary Outcome: Number of Participants With Family Practitioner Visits in Past 6 Months- Primary Analysis
Description: Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Participants | 102 | 979
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Test type: Other; p = 0.758, Chi-squared

26. Primary Outcome: Mean Number of Family Practitioner Visits in Past 6 Months- Primary Analysis
Description: Mean number of family practitioner visits within the last six months due to any cause among those who had at least 1 family practitioner visit is reported in this outcome measure. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 21
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Family Practitioner Visits
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 102 | 979
Family Practitioner Visits | 2 (1.2) | 2 (2)
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Test type: Other; p = 0.616, t-test, 2 sided

27. Primary Outcome: Number of Participants With Cardiologist Visits in Past 6 Month- Primary Analysis
Description: Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Participants | 21 | 130
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Test type: Other; p = 0.086, Chi-squared

28. Primary Outcome: Mean Number of Cardiologist Visits in Past 6 Months- Primary Analysis
Description: Mean number of cardiologist visits within the last six months due to any cause among those who had at least 1 cardiologist visit is reported in this outcome measure. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 21
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Cardiologist Visits
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 21 | 130
Cardiologist Visits | 1.6 (1.2) | 1.8 (1.5)
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Test type: Other; p = 0.528, t-test, 2 sided

29. Primary Outcome: Number of Participants With Neurologist Visits in Past 6 Months - Primary Analysis
Description: Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: 6 months before the survey was taken, during 1 year of data identification (Year 2023); available retrospective data was evaluated over approximately 1.41 month of this observational study.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Participants | 72 | 374
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Test type: Other; p < 0.001, Chi-squared

30. Primary Outcome: Mean Number of Neurologist Visits in Past 6 Months- Primary Analysis
Description: Mean number of neurologist visits within the last six months due to any cause among those who had at least 1 neurologist visit is reported in this outcome measure. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 21
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Neurologist Visits
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 72 | 374
Neurologist Visits | 2.6 (6) | 2 (1.3)
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Test type: Other; p = 0.395, t-test, 2 sided

31. Primary Outcome: Number of Participants With Traditional Healthcare Provider Visits in Past 6 Months- Primary Analysis
Description: Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 135 | 1260
Participants | 132 | 1228
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Test type: Other; p = 1, Chi-squared

32. Primary Outcome: Mean Number of Traditional Healthcare Provider Visits in Past 6 Months- Primary Analysis
Description: Mean number of traditional healthcare provider visits within the last six months due to due to any cause among those who had at least 1 healthcare provider visit is reported in this outcome measure. Analysis was performed using IPTW method to adjust for confounding by the covariate.
Time Frame: as for outcome 21
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Traditional Healthcare Provider Visits
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 132 | 1228
Traditional Healthcare Provider Visits | 9.5 (10.6) | 7.8 (8.1)
Statistical Analysis 1: Comparison: Rimegepant vs Triptans; Test type: Other; p = 0.08, t-test, 2 sided

33. Secondary Outcome: Research and Development (RAND-36) Physical Component Score, Mental Component Score and Global Health Score - Sensitivity Analysis.
Description: as for outcome 12
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in the study. For sensitivity analysis a subset of rimegepant users with less than 12 days of rimegepant use per month were included and the numbers were adjusted using IPTW method, which created pseudo population, leading to difference from the sample sizes before IPTW.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Rimegepant (Users With <12 Days of Use): Participants who were acute rimegepant users with days of use < 12 days per month for migraine at the time of survey (NHWS in Year 2023) were included. No intervention was administered as a part of this study.
- Triptans: Participants who responded to use triptans orally for migraine at the time of survey (NHWS in Year 2023) were included. No intervention was administered as a part of this study.
Arm/Group | Rimegepant (Users With <12 Days of Use) | Triptans
Number analyzed (Participants) | 103 | 1257
Units on a scale
  Mental summary composite T score | 39.1 (11.9) | 38.1 (12.4)
  Physical summary composite T score | 40.6 (11.5) | 41.2 (11.6)
  Global health composite T score | 38.3 (12) | 38 (12.4)
Statistical Analysis 1: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Mental summary composite T score; Test type: Other; p = 0.426, t-test, 2 sided
Statistical Analysis 2: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Physical summary composite T score; Test type: Other; p = 0.602, t-test, 2 sided
Statistical Analysis 3: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Global health composite T score; Test type: Other; p = 0.815, t-test, 2 sided

34. Secondary Outcome: European Quality of Life 5 Dimensions 5 Level (EQ-5D-5L) Index Score- Sensitivity Analysis
Description: as for outcome 13
Time Frame: as for outcome 1
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rimegepant (Users With <12 Days of Use) | Triptans
Number analyzed (Participants) | 103 | 1257
Units on a scale | 0.8 (0.2) | 0.7 (0.2)
Statistical Analysis 1: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Test type: Other; p = 0.189, t-test, 2 sided

35. Secondary Outcome: EQ-5D-5L Visual Analog Scale (VAS) Score- Sensitivity Analysis
Description: as for outcome 14
Time Frame: as for outcome 1
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rimegepant (Users With <12 Days of Use) | Triptans
Number analyzed (Participants) | 103 | 1257
Units on a scale | 69.6 (20.2) | 68.9 (19.5)
Statistical Analysis 1: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Test type: Other; p = 0.727, t-test, 2 sided

36. Secondary Outcome: Percentage of Work Time Missed in Past 7 Days Based on Work Productivity and Activity Impairment - General Health (WPAI-GH) Questionnaire- Sensitivity Analysis
Description: The WPAI is a standardized PRO that assessed the previous 7 days of completing the questionnaire. WPAI:GH is a self-reported measure of work productivity and impairment, which had four scores: absenteeism (work time missed); presenteeism (impairment at work/reduced on the job effectiveness); work productivity loss (overall work impairment/absenteeism plus presenteeism); and total activity impairment. The scores for percentage of work time missed ranged from 0 (no impairment/high productivity) to 100% (high impairment/total loss of work productivity) with higher score indicating greater impairment and less productivity. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 15
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: Percentage work time missed
Arm/Group | Rimegepant (Users With <12 Days of Use) | Triptans
Number analyzed (Participants) | 103 | 1257
Percentage work time missed | 6.4 (14) | 8.8 (19.2)
Statistical Analysis 1: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Test type: Other; p = 0.237, t-test, 2 sided

37. Secondary Outcome: Percentage Impairment Experienced While at Work in Past 7 Days Based on WPAI-GH Questionnaire-Sensitivity Analysis
Description: The WPAI is a standardized PRO that assessed the previous 7 days of completing the questionnaire. WPAI:GH is a self-reported measure of work productivity and impairment, which had four scores: absenteeism (work time missed); presenteeism (impairment at work/reduced on the job effectiveness); work productivity loss (overall work impairment/absenteeism plus presenteeism); and total activity impairment. The scores for percentage impairment experienced ranged from 0 (no impairment/high productivity) to 100% (high impairment/total loss of work productivity) with higher score indicating greater impairment and less productivity. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 15
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: Percentage impairment
Arm/Group | Rimegepant (Users With <12 Days of Use) | Triptans
Number analyzed (Participants) | 103 | 1257
Percentage impairment | 28.1 (26.4) | 25 (24.7)
Statistical Analysis 1: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Test type: Other; p = 0.401, t-test, 2 sided

38. Secondary Outcome: Percentage Overall Work Impairment in Past 7 Days Based on WPAI-GH Questionnaire- Sensitivity Analysis
Description: The WPAI is a standardized PRO that assessed the previous 7 days of completing the questionnaire. WPAI:GH is a self-reported measure of work productivity and impairment, which had four scores: absenteeism (work time missed); presenteeism (impairment at work/reduced on the job effectiveness); work productivity loss (overall work impairment/absenteeism plus presenteeism); and total activity impairment. The scores for percentage overall work impairment experienced ranged from 0 (no impairment/high productivity) to 100% (high impairment/total loss of work productivity) with higher score indicating greater impairment and less productivity. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 15
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: Percentage work impairment
Arm/Group | Rimegepant (Users With <12 Days of Use) | Triptans
Number analyzed (Participants) | 103 | 1257
Percentage work impairment | 30.4 (28.5) | 28.4 (27.9)
Statistical Analysis 1: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Test type: Other; p = 0.609, t-test, 2 sided

39. Secondary Outcome: Percentage Total Activity Impairment in Past 7 Days Based on WPAI-GH Questionnaire- Sensitivity Analysis
Description: The WPAI is a standardized PRO that assessed the previous 7 days of completing the questionnaire. WPAI:GH is a self-reported measure of work productivity and impairment, which had four scores: absenteeism (work time missed); presenteeism (impairment at work/reduced on the job effectiveness); work productivity loss (overall work impairment/absenteeism plus presenteeism); and total activity impairment. The scores for percentage of total activity impairment ranged from 0 (no impairment/high productivity) to100% (high impairment/total loss of work productivity) with higher score indicating greater impairment and less productivity. In this outcome measure, percentage total activity impairment among total population, employed, unemployed and disabled is reported. Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 15
Population: Analysis population included all eligible participants whose data were retrieved and observed in the study. For sensitivity analysis a subset of rimegepant users with less than 12 days of rimegepant use per month were included and the numbers were adjusted using IPTW method, which created pseudo population, leading to difference from the sample sizes before IPTW. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage activity impairment
Arm/Group | Rimegepant (Users With <12 Days of Use) | Triptans
Number analyzed (Participants) | 103 | 1257
Percentage activity impairment
  Total activity impairment | 37.6 (28) | 34.4 (28.3)
  Activity impairment among employed: number analyzed (Participants) | 63 | 782
  Activity impairment among employed | 30.6 (25.6) | 28.3 (25.9)
  Activity impairment among unemployed: number analyzed (Participants) | 31 | 383
  Activity impairment among unemployed | 44.4 (27.7) | 38.7 (28.3)
  Activity impairment among disabled: number analyzed (Participants) | 9 | 92
  Activity impairment among disabled | 63.3 (26.9) | 68.8 (19.3)
Statistical Analysis 1: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Total activity impairment; Test type: Other; p = 0.265, t-test, 2 sided
Statistical Analysis 2: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Activity impairment among employed; Test type: Other; p = 0.496, t-test, 2 sided
Statistical Analysis 3: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Activity impairment among unemployed; Test type: Other; p = 0.268, t-test, 2 sided
Statistical Analysis 4: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Activity impairment among disabled; Test type: Other; p = 0.57, t-test, 2 sided

40. Secondary Outcome: Migraine Disability Assessment Scale (MIDAS) Total Score and Individual Item Scores- Sensitivity Analysis
Description: as for outcome 19
Time Frame: as for outcome 19
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rimegepant (Users With <12 Days of Use) | Triptans
Number analyzed (Participants) | 103 | 1257
Units on a scale
  MIDAS (Total score) | 25.6 (36) | 21.6 (29.1)
  MIDAS Item 1 (MGMIDAS1) | 1.9 (5.8) | 1.8 (4.9)
  MIDAS Item 2 (MGMIDAS2) | 4.9 (9.3) | 4.1 (7.6)
  MIDAS Item 3 (MGMIDAS3) | 7.8 (12.1) | 5.8 (7.8)
  MIDAS Item 4 (MGMIDAS4) | 7 (9.8) | 6.1 (8.6)
  MIDAS Item 5 (MGMIDAS5) | 4.1 (7.7) | 3.8 (8.1)
  MIDAS Item 6 (MGMIDAS6) | 19.5 (21.9) | 14.3 (16.8)
  MIDAS Item 7 (MGMIDAS7) | 6.7 (1.8) | 6.7 (1.9)
Statistical Analysis 1: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; MIDAS (Total score); Test type: Other; p = 0.266, t-test, 2 sided
Statistical Analysis 2: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; MIDAS Item 1 (MGMIDAS1); Test type: Other; p = 0.884, t-test, 2 sided
Statistical Analysis 3: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; MIDAS Item 2 (MGMIDAS2); Test type: Other; p = 0.373, t-test, 2 sided
Statistical Analysis 4: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; MIDAS Item 3 (MGMIDAS3); Test type: Other; p = 0.109, t-test, 2 sided
Statistical Analysis 5: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; MIDAS Item 4 (MGMIDAS4); Test type: Other; p = 0.368, t-test, 2 sided
Statistical Analysis 6: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; MIDAS Item 5 (MGMIDAS5); Test type: Other; p = 0.714, t-test, 2 sided
Statistical Analysis 7: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; MIDAS Item 6 (MGMIDAS6); Test type: Other; p = 0.020, t-test, 2 sided
Statistical Analysis 8: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; MIDAS Item 7 (MGMIDAS7); Test type: Other; p = 0.889, t-test, 2 sided

41. Secondary Outcome: Number of Participants According to MIDAS Grade - Sensitivity Analysis
Description: as for outcome 20
Time Frame: as for outcome 19
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant (Users With <12 Days of Use) | Triptans
Number analyzed (Participants) | 103 | 1257
Participants
  MIDAS Grade I | 29 | 398
  MIDAS Grade II | 17 | 159
  MIDAS Grade III | 23 | 270
  MIDAS Grade IV | 34 | 430
Statistical Analysis 1: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; MIDAS Grade I to Grade IV; Test type: Other; p = 0.675, Chi-squared

42. Secondary Outcome: Number of Participants With Emergency Room (ER) Visits in Past 6 Months- Sensitivity Analysis
Description: Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 21
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant (Users With <12 Days of Use) | Triptans
Number analyzed (Participants) | 103 | 1257
Participants | 27 | 301
Statistical Analysis 1: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Test type: Other; p = 0.651, Chi-squared

43. Secondary Outcome: Number of ER Visits in Past 6 Months- Sensitivity Analysis
Description: as for outcome 22
Time Frame: as for outcome 21
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: ER visits
Arm/Group | Rimegepant (Users With <12 Days of Use) | Triptans
Number analyzed (Participants) | 27 | 301
ER visits | 1.4 (0.6) | 1.8 (1.5)
Statistical Analysis 1: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Test type: Other; p = 0.004, t-test, 2 sided

44. Secondary Outcome: Number of Participants With Hospitalizations in Past 6 Months- Sensitivity Analysis
Description: Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 21
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant (Users With <12 Days of Use) | Triptans
Number analyzed (Participants) | 103 | 1257
Participants | 11 | 111
Statistical Analysis 1: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Test type: Other; p = 0.477, Chi-squared

45. Secondary Outcome: Mean Number of Hospitalizations in Past 6 Months- Sensitivity Analysis
Description: as for outcome 24
Time Frame: as for outcome 21
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: Hospitalizations
Arm/Group | Rimegepant (Users With <12 Days of Use) | Triptans
Number analyzed (Participants) | 11 | 111
Hospitalizations | 1.2 (0.4) | 1.8 (1.3)
Statistical Analysis 1: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Test type: Other; p = 0.002, t-test, 2 sided

46. Secondary Outcome: Number of Participants With Family Practitioner Visits in Past 6 Months- Sensitivity Analysis
Description: Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 21
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant (Users With <12 Days of Use) | Triptans
Number analyzed (Participants) | 103 | 1257
Participants | 76 | 976
Statistical Analysis 1: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Test type: Other; p = 0.555, Chi-squared

47. Secondary Outcome: Mean Number of Family Practitioner Visits in Past 6 Months- Sensitivity Analysis
Description: as for outcome 26
Time Frame: as for outcome 21
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: Family Practitioner Visits
Arm/Group | Rimegepant (Users With <12 Days of Use) | Triptans
Number analyzed (Participants) | 76 | 976
Family Practitioner Visits | 1.9 (1.2) | 2 (1.9)
Statistical Analysis 1: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Test type: Other; p = 0.371, t-test, 2 sided

48. Secondary Outcome: Number of Participants With Cardiologist Visits in Past 6 Months- Sensitivity Analysis
Description: Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 21
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant (Users With <12 Days of Use) | Triptans
Number analyzed (Participants) | 103 | 1257
Participants | 14 | 137
Statistical Analysis 1: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Test type: Other; p = 0.501, Chi-squared

49. Secondary Outcome: Mean Number of Cardiologist Visits in Past 6 Months- Sensitivity Analysis
Description: as for outcome 28
Time Frame: as for outcome 21
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: Cardiologist Visits
Arm/Group | Rimegepant (Users With <12 Days of Use) | Triptans
Number analyzed (Participants) | 14 | 137
Cardiologist Visits | 1.3 (0.5) | 1.7 (1.4)
Statistical Analysis 1: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Test type: Other; p = 0.014, t-test, 2 sided

50. Secondary Outcome: Number of Participants With Neurologist Visits in Past 6 Months- Sensitivity Analysis
Description: Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 29
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant (Users With <12 Days of Use) | Triptans
Number analyzed (Participants) | 103 | 1257
Participants | 57 | 358
Statistical Analysis 1: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Test type: Other; p < 0.001, Chi-squared

51. Secondary Outcome: Mean Number of Neurologist Visits in Past 6 Months- Sensitivity Analysis
Description: as for outcome 30
Time Frame: as for outcome 21
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: Neurologist Visits
Arm/Group | Rimegepant (Users With <12 Days of Use) | Triptans
Number analyzed (Participants) | 57 | 358
Neurologist Visits | 2.6 (6.4) | 1.9 (1.3)
Statistical Analysis 1: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Test type: Other; p = 0.392, t-test, 2 sided

52. Secondary Outcome: Number of Participants With Traditional Healthcare Provider Visits in Past 6 Months- Sensitivity Analysis
Description: Analysis was performed using IPTW method to adjust for confounding by the covariates.
Time Frame: as for outcome 21
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant (Users With <12 Days of Use) | Triptans
Number analyzed (Participants) | 103 | 1257
Participants | 101 | 1227
Statistical Analysis 1: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Test type: Other; p = 1, Chi-squared

53. Secondary Outcome: Mean Number of Traditional Healthcare Provider Visits in Past 6 Months- Sensitivity Analysis
Description: as for outcome 32
Time Frame: as for outcome 21
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: Traditional Healthcare Provider Visits
Arm/Group | Rimegepant (Users With <12 Days of Use) | Triptans
Number analyzed (Participants) | 101 | 1227
Traditional Healthcare Provider Visits | 9.2 (10.3) | 7.7 (8)
Statistical Analysis 1: Comparison: Rimegepant (Users With <12 Days of Use) vs Triptans; Test type: Other; p = 0.143, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events and all-cause mortality were not planned to be evaluated/ monitored for the study.
Description: Due to non-interventional nature of the study and nature of data sources, the minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) could not be met, hence adverse events and all-cause mortality were not planned to be assessed or monitored (thus at risk appears "0").
Groups:
- Rimegepant: Participants with self-reported diagnosis of migraine currently on rimegepant use at the time of survey completion (NHWS in year 2023) were included. No intervention was administerred as part of this study.
- Triptans: Participants with self-reported diagnosis of migraine currently on triptan use at the time of survey completion (NHWS in year 2023) were included. No intervention was administerred as part of this study.
Arm/Group | Rimegepant | Triptans
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT06680206/Prot_SAP_000.pdf